CLINICAL TRIAL: NCT02087098
Title: Czech Observational Study to Evaluate Quality of Life in Patients Switched to Vesicare™ (Solifenacin) From Other Antimuscarinics
Brief Title: A Study to Evaluate Quality of Life in Patients Switched to Solifenacin From Other Antimuscarinics
Acronym: VEST
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: VEST-001
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Bladder, Overactive
Keywords: overactive bladder; solifenacin; quality of life
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with residual OAB symptoms: Urge urinary incontinence, urgency, and frequency after treatment with other antimuscarinics
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Solifenacin — Patients with residual OAB symptoms (urge urinary incontinence, urgency, and frequency) after treatment with other antimuscarinics
  Other Names: Vesicare

SUMMARY:
This is a 12 month non-interventional study with solifenacin succinate, evaluating the effect of solifenacin on quality of life (QoL) of patients previously treated with antimuscarinics (Males and Females with Overactive Bladder (OAB) symptoms withdrawing their treatment with antimuscarinics because of safety and/or efficacy reasons) - measured by Perception of Treatment Satisfaction (TS-VAS) and to evaluate the effect of solifenacin on quality of life measured by Over Active Bladder-q Short Form (OAB-q SF), EuroQol Group scoring system (EQ-5D-5L).

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to complete the questionnaires
* Diagnosis of OAB
* Previous unsuccessful OAB medication (antimuscarinic treatment for at least 1 month) less than 4 weeks ago defined by:

  * number of micturitions > 8/24 h or
  * decrease in urgency urinary incontinence (UUI) or incontinence episodes / 24 h less than 50% or
  * decrease in urgency episodes / 24 h less than 50% or
  * decrease in number of micturitions / 24 h less than 20% or
  * not acceptable tolerability
* Eligible to start Vesicare™ 5 or 10 mg according to Summary of Product Characteristics (SmPC)

Exclusion Criteria:

* History of stress incontinence
* Active urinary tract infection (confirmed by positive urine analysis)
* Symptoms suggestive of severe Bladder Outlet Obstruction (BOO) defined as Peak urinary flow rate (Qmax) < 10ml/sc and/or Postvoid residual urine volume (PVR) > 150 ml
* Uncontrolled Diabetes Mellitus
* History of drug and/or alcohol abuse at the time of enrolment
* History of acute urinary retention, severe gastrointestinal obstruction (including paralytic ileus or intestinal atony or toxic megacolon or severe ulcerative colitis), myasthenia gravis, uncontrolled narrow glaucoma or swallow anterior chamber or deemed to be at risk for these conditions.
* Undergoing hemodialysis or has severe renal impairment or moderate hepatic impairment and who are on treatment with a potent CYP3A4 inhibitor
* Previous treatment with solifenacin
* Likely to participate in another study during study period of 12 months from study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OAB symptoms being treated by urologists in Czech Republic
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Over Active Bladder questionnaire Short Form (OAB-q SF) score | baseline, month 6 and 12
Change from baseline of Patient Assessment of Treatment Satisfaction (TS-VAS) | baseline, month 6 and 12
Change from baseline in EuroQol Group system (EQ-5D-5L) score | baseline, month 6 and 12

SECONDARY OUTCOMES:
Change in QoL according to previous antimuscarinic treatment and sex (assessed by: TS-VAS score, OAB-q SF score, EQ-5D-5L) | baseline, month 1, 3, 6 and 12
Change from baseline in OAB symptoms assessed by micturition diary | baseline, month 1, 3, 6 and 12
  Mean number of urgency episode per 24 hours, mean number of micturition per 24 hours, mean number of nocturia episodes per 24 hours, mean number of urge incontinence (UUI) episodes per week
Persistence to therapy (measured by proportion of Days Covered (PDC, threshold of 80 percent during the measurement period), median length of therapy (days)) | 12 months
Occurence of adverse drug reaction | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (60):
- Czechia (60):
  - Site CZ42003 Private Practice, Benešov
  - Site CZ42001 Private Practice, Beroun
  - Site CZ42014 Private Practice, Blansko
  - Site CZ42023 Private Practice, Boskovice
  - Site CZ42032 Private Practice, Brno
  - Site CZ42034 Hospital, Brno
  - Site CZ42035 Private Practice, Brno
  - Site CZ42036 Private Practice, Brno
  - Site CZ42038 Private Practice, Brno
  - Site CZ42039 Private Practice, Brno
  - Site CZ42058 Hospital, Brno
  - Site CZ42059 Hospital, Brno
  - Site CZ42025 Private Practice, Cheb
  - Site CZ42048 Private Practice, Dvůr Králové
  - Site CZ42040 Private Practice, Havlíčkův Brod
  - Site CZ42015 Private Practice, Hodonín
  - Site CZ42045 Private Practice, Hradec Králové
  - Site CZ42051 Private Practice, Jičín
  - Site CZ42027 Private Practice, Jindřichŭv Hradec
  - Site CZ42029 Private Practice, Jindřichŭv Hradec
  - Site CZ42026 Private Practice, Karlovy Vary
  - Site CZ42028 Private Practice, Karlovy Vary
  - Site CZ42030 Private Practice, Klatovy
  - Site CZ42049 Private Practice, Litoměřice
  - Site CZ42021 Private Practice, Litovel
  - Site CZ42050 Private Practice, Most
  - Site CZ42054 Private Practice, Ostrava
  - Site CZ42055 Private Practice, Ostrava
  - Site CZ42056 Private Practice, Ostrava
  - Site CZ42057 Private Practice, Ostrava
  - Site CZ42005 Private Practice, Pardubice
  - Site CZ42008 Private Practice, Pardubice
  - Site CZ42024 Private Practice, Pilsen
  - Site CZ42002 Private Practice, Prague
  - Site CZ42004 Private Practice, Prague
  - Site CZ42006 Private Practice, Prague
  - Site CZ42007 Private Practice, Prague
  - Site CZ42009 Private Practice, Prague
  - Site CZ42010 Private Practice, Prague
  - Site CZ42011 Private Practice, Prague
  - Site CZ42060 Private Practice, Prague
  - Site CZ42044 Private Practice, Roudnice nad Labem
  - Site CZ42031 Private Practice, Strakonice
  - Site CZ42020 Private Practice, Svitavy
  - Site CZ42047 Private Practice, Teplice
  - Site CZ42053 Private Practice, Teplice
  - Site CZ42042 Private Practice, Trutnov
  - Site CZ42052 Private Practice, Turnov
  - Site CZ42018 Hospital, Uherské Hradiště
  - Site CZ42019 Private Practice, Uherské Hradiště
  - Site CZ42043 Private Practice, Ústí nad Labem
  - Site CZ42046 Private Practice, Ústí nad Labem
  - Site CZ42041 Hospital, Velké Meziříčí
  - Site CZ42016 Private Practice, Vsetín
  - Site CZ42017 Private Practice, Vsetín
  - Site CZ42012 Private Practice, Zlín
  - Site CZ42013 Private Practice, Zlín
  - Site CZ42022 Private Practice, Zlín
  - Site CZ42033 Private Practice, Znojmo
  - Site CZ42037 Hospital, Znojmo